CLINICAL TRIAL: NCT05797285
Title: A Randomized Clinical Pilot Evaluating The Efficacy For Two Application Regimens Of A Unique Keratin Based Graft In The Treatment Of Non-Healing Diabetic Foot Ulcers
Brief Title: Evaluating The Efficacy Of A Keratin Graft In Treating Non-Healing Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProgenaCare Global, LLC (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRG-PM-DFU-01
Record Dates: First submitted 2023-03-09; First posted 2023-04-04 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Ulcer Healing; Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Wound Care
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: In this trial, two groups of subjects with diabetic foot ulcers (DFUs), will receive standard of care (SOC) treatment for their condition. The study has two phases: a 14-day screening phase to determine eligibility, and a 13-week treatment phase. Half of the patients will be randomized to a 510K FDA cleared ProgenaMatrix applied weekly and the other half will be randomized to a 510K FDA cleared ProgenaMatrix applied bi-weekly (i.e., once every two weeks).
  SOC includes offloading the DFU with controlled ankle movement (CAM) boots or total contact casting, appropriate sharp or surgical debridement, and wound care covering with ProgenaMatrix followed by a padded 3-layer dressing of 4x4 gauze, soft roll, and compressive wrap.
Masking Description: The treatments in this study will not be masked. Assessment of the primary study objective (wound closure) will be overseen by an adjudication panel of at least two wound care experts to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Weekly Human Keratin Graft Application (Experimental): Patients randomized into this arm will receive standard of care (offloading, debridement, and three-layer outer dressing) with the test material, the human keratin graft, reapplied weekly to the target wound.
  Interventions: Device: human keratin graft
- Bi-Weekly Human Keratin Graft Application (Experimental): Patients randomized into this arm will receive standard of care (offloading, debridement, and three-layer outer dressing) with the test material, the human keratin graft, reapplied every other week to the target wound.
  Interventions: Device: human keratin graft

INTERVENTIONS:
Device: human keratin graft — The intervention to be applied is an advanced wound care matrix composed of human keratin to be applied at two different treatment frequencies.
  Other Names: ProgenaMatrix

SUMMARY:
The goal of this clinical pilot is to collect patient outcome data on a commercially available, keratin-based skin substitute matrix: ProgenaMatrix®. In this trial, two groups of patients with diabetic foot ulcers (DFUs) will be randomized to receive treatment with ProgenaMatrix applied either weekly or bi-weekly to the target wound. Researchers will compare how weekly or bi-weekly application of ProgenaMatrix affects the healing of DFUs.

The primary questions to be answered are:

1. How many patients achieve wound closure in 12 weeks with ProgenaMatrix treatment? And
2. What is the change in wound area during the trial in each group?

DETAILED DESCRIPTION:
ProgenaMatrix® is a human keratin graft that is 510K approved for application on diabetic foot wounds and has been shown in case studies and clinical practice to assist in wound healing . Additionally, a study published by Tang and Kirsner showed that keratin stimulates human keratinocyte migration and types IV and VII collagen expression. Therefore, based on this early promising data, a larger pilot is necessary to further validate these results and identify the likelihood of wound healing with weekly versus bi-weekly application. For consistency, one type of wound will be studied in this trial and DFU's have been chosen as they are some of the most common wounds seen in the wound clinics.

The purpose of this clinical evaluation is to collect patient outcome data on a commercially available 510K FDA cleared synthetic, absorbable skin substitute matrix. The commercially available product is ProgenaMatrix® Advanced Wound Graft and consists of Human Keratin Matrix. In this trial, two groups of subjects with diabetic foot ulcers (DFUs), will receive standard of care (SOC) treatment for their condition. Half of the patients will be randomized to a 510K FDA cleared ProgenaMatrix® applied weekly and the other half will be randomized to a 510K FDA cleared ProgenaMatrix® applied bi-weekly (i.e., once every two weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or 2 diabetes mellitus
* Target diabetic foot ulcer with a minimum surface area of 1.0 cm^2 and a maximum surface area of 20.0 cm^2 measured post-debridement with photographic planimetry.
* Target ulcer must have been present for a minimum of 4 weeks and maximum of 52 weeks of standard of care prior to initial screening
* Target ulcer must be located on the foot with at least 50% of its area below the malleolus
* Target ulcer must be full thickness on the foot or ankle that does not probe to bone
* Adequate circulation in the affected foot documented within 3 months of initial screening visit, as determined by one of the following: transcutaneous oximetry measurement (TCOM) greater or equal to 30 mmHg, ankle-brachial index (ABI) between 0.7 and 1.3, biphasic pulse volume recording (PVR), toe-brachial index (TBI) greater than 0.6, or arterial Doppler ultrasound evaluating for biphasic dorsalis pedis and posterior tibial vessels at the ankle level
* If subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer
* Target ulcers on the plantar aspect of the foot must be offloaded for at least 14 days prior to randomization
* Subject must consent to using the prescribed off-loading method for the duration of the study
* Subject must agree to attend weekly study visits required by the protocol
* Subject must be willing and able to participate in the informed consent process

Exclusion Criteria:

* Subjects known to have a life expectancy of < 6 months
* Infection of the target ulcer or cellulitis in the surrounding skin
* Presence of osteomyelitis or exposed bone, or wounds that probe to bone or joint capsule on investigator's exam or radiographic evidence
* Infection in the target ulcer requiring systemic antibiotic therapy
* Subjects receiving immunosuppressants (including systemic corticosteroids > 10 mg Prednisone per day or equivalent) or cytotoxic chemotherapy
* Topical application of steroids to the ulcer surface within one month of initial screening
* Subjects with previous partial amputation on the affected foot that impedes proper offloading of the target ulcer
* Subjects with a glycated hemoglobin (HbA1c) greater than or equal to 13% taken at or within 3 months of the initial screening visit
* Subjects with a serum creatinine level ≥ 3.0mg/dL within 6 months of randomization
* Surface area of the target ulcer reduces in size by more than 30% in the two weeks between the initial screening and randomization during which they are subject to standard of care
* Subjects with acute or inactive Charcot foot that impedes proper offloading of the target ulcer
* Women who are pregnant or considering becoming pregnant within the next 6 months
* Subjects with end stage renal disease requiring dialysis
* Subjects who participated in a clinical trial involving treatment with an investigational product within the previous 30 days
* Subjects who, in the opinion of the investigator, have a medical or psychological condition that may interfere with study assessments
* Subjects treated with hyperbaric oxygen therapy or a cellular and/or tissue product (CTP) in the 30 days prior to the initial screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 12 weeks
  The proportion of subjects that achieve complete closure of the target wound with each treatment.

SECONDARY OUTCOMES:
Time to Wound Closure | From date of randomization until date of documented wound closure, assessed up to 12 weeks
  The time required for target ulcers to achieve complete closure with each treatment.
Wound Area Change | From date of randomization until date of documented wound closure or study conclusion, whichever comes first, assessed up to 12 weeks
  The change in target wound area between treatment visits.
Change in Peripheral Neuropathy | From date of randomization until date of documented wound closure or study conclusion, whichever comes first, assessed up to 12 weeks
  Changes in peripheral neuropathy of the foot with the target ulcer between treatment visits, assessed by the standard 10-point Semmes-Weinstein monofilament exam.
Change in Wound Pain | From date of randomization until date of documented wound closure or study conclusion, whichever comes first, assessed up to 12 weeks
  Changes in pain in the target ulcer assessed by the numerical pain rating scale from 0 (no pain) to 10 (worst pain possible).
Change in Quality of Life | From date of first screening until date of documented wound closure or study conclusion, whichever comes first, assessed up to 15 weeks
  Changes in patient quality of life relating to their wound using the wound quality of life assessment with 17 questions answered on a scale of 0 ("not at all") to 4 ("very much").

OTHER OUTCOMES:
Presence of Cellulitis and Infection | 12 weeks
  Difference in number of participants presenting with cellulitis and/or infection in or around the target ulcer between treatment groups.
Number of Adverse Events Observed | 15 weeks
  The number and type of adverse events observed during the study.

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM,MD,PhD, Study Chair — University of Southern California
Locations (3):
- United States (3):
  - Doctors Research Network, Miami, Florida
  - Foot and Ankle Specialists of the Mid-Atlantic (FASMA), Frederick, Maryland
  - Foot and Ankle Specialists of the Mid-Atlantic (FASMA), Salem, Virginia

IPD SHARING:
Plan to Share IPD: Undecided